CLINICAL TRIAL: NCT02519270
Title: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Intravenous Doses of IGN002 Administered Weekly to Subjects With Refractory Non-Hodgkin Lymphoma (NHL)
Brief Title: Phase 1, Dose-Escalation Study of IGN002 in NHL Subjects
Acronym: NHL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Reasons
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGN002-101
Record Dates: First submitted 2015-08-03; First posted 2015-08-10 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation Stage/ Expansion Stage (Experimental): The Dose-Escalation Stage will employ a modified 3 + 3 cohort design, subjects will receive up to 26 doses of IGN002.
  In the Expansion Stage, subjects will receive up to 24 doses of IGN002 at the maximum tolerated dose administered weekly in three 8-week cycles.
  Interventions: Biological: IGN002

INTERVENTIONS:
Biological: IGN002 — IGN002 is a monoclonal antibody fusion protein.

SUMMARY:
A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Intravenous Doses of IGN002 Administered Weekly to Subjects with Refractory Non-Hodgkin Lymphoma (NHL)

DETAILED DESCRIPTION:
This open-label, non-randomized, first-in-human Phase 1 study involves two stages:

In the Dose-Escalation Stage, ascending dose cohorts will be treated in 2 periods until the maximum tolerated dose is identified. In Period 1, subjects will receive 2 doses of IGN002 administered weekly. In Period 2, subjects will receive up to 24 additional doses of IGN002 administered weekly in three 8-week cycles. Subjects that have not progressed following the treatment period will be followed for another 6 months.

In the Expansion Stage, subjects will receive up to 24 doses of IGN002 at the identified maximum tolerated dose administered weekly in three 8-week cycles. Subjects that have not progressed following the treatment period will be followed for another 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of immunohistochemistry (IHC)-confirmed CD20-positive (with no subsequent history of CD20-negativity) B-cell, NHL, including diffuse large B cell (DLBCL), mantle cell, marginal zone, lymphoplasmacytic, follicular, transformed follicular, or primary mediastinal B cell lymphoma
* Refractory disease, having failed available therapies
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy > 3 months
* Adequate organ function

Exclusion Criteria:

* Treatment with an approved or investigational chemotherapy drug within 28 days of Day 1
* Treatment with an approved or investigational anti-CD20 drug within 28 days of Day 1
* Treatment with an approved or investigational biologic drug that does not target CD20 within 90 days of Day 1
* Radiation therapy within 4 weeks of Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple doses of IGN002 administered weekly as an intravenous (IV) infusion to subjects with refractory NHL | Weekly for 6 months
  Adverse Event collection and assessment will be done for all potentially treated subjects to assess the safety, tolerability, and determine the maximum tolerated dose

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (PK) profile of ascending doses of IGN002 administered weekly | Weekly for 6 months
  Pharmacokinetic (PK) parameters such as Maximum concentration (Cmax), time to maximum concentration (Tmax), minimum concentration(Cmin), area under the curve (AUC), half-life (t1/2), clearance (CL)
To assess the anti-tumor activity of IGN002 using the Lugano Classification for NHL | Every 8 weeks for 6 months, then at 1, 3 and 6 months
  Determine the therapeutic effects, in terms of objective response rate and duration, of the therapeutic agent in NHL patients.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA, Santa Monica, California
  - UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No